CLINICAL TRIAL: NCT06806020
Title: Effect Of Scientific Exercise Approach For Scoliosis Versus Barcelona Scoliosis Physical Therapy School On Correction Of Adolescent Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Huda Hashad, huda mohamed hashad, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KFSIRB200-404
Record Dates: First submitted 2025-01-27; First posted 2025-02-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Scoliosis; Idiopathic Scoliosis; Adolescent Scoliosis
Keywords: idiopathic adolescent scoliosis SEAS BSPTS; SEAS approach; BSPTS
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Intervention Model Description: Intervention study model Parallel assignment The study will include 30 adolescent idiopathic scoliosis patients ( age12-16 years old ) subjects meeting the inclusion criteria will be randomly assigned to two experimental groups : First experimental group: children in this group will receive BSPTS school Second experimental group: children in this group will receive SEAS approach
Masking Description: Intervention study model Parallel assignment The study will include 30 idiopathic adolescent scoliosis patients( age 12-16 years old ) subjects meeting the inclusion criteria will be randomly assigned to two experimental groups : First experimental group: children in this group will receive BSPTS school training Second experimental group: children in this group will receive SEAS approach training
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group (1) (Experimental): SEAS approach
  Interventions: Other: SEAS approach
- group (2) (Experimental): BSPTS school
  Interventions: Other: BSPTS school

INTERVENTIONS:
Other: SEAS approach — The SEAS approach provides a thorough evaluation of the patient before the treatment starts. In addition to the usual measurements for the specific assessment of the scoliosis (Cobb degrees, Bunnel, trunk decompensation, sagittal postural structure and aesthetic parameters), the patient performs a series of tests. The objectives are: assessment of physical conditions (strength and elasticity of certain muscle areas that are more likely 6 influence the structure of the pelvis and the spine), assessment of neuromotor ability related to the alignment of the spine and the pelvis (balance, management of body movements with closed eyes, optical/manual skills) (Romano et al, 2015).
  The main aim of SEAS is to reverse the Stokes vicious cycle, so, the abnormal loading created by the scoliosis with an asymmetric growth leading to worsening of curves that will lead to further asymmetric growth due to increased asymmetrical loading (ettany et al 2014).
  The goal of SEAS exercises is to develop an a
  Arms: group (1)
Other: BSPTS school — Barcelona scoliosis physical therapy school (BSPTS): Based on the theory that scoliosis posture promotes curve progression, according to the "vicious cycle" model, Barcelona Scoliosis Physical Therapy School (BSPTS) is a physiotherapeutic method that can be defined as a therapy plan of cognitive, sensory-motor, and kinesthetic training to teach the patient to improve their scoliosis 3D posture and shape. The BSTPS method aims to: 1) improve aesthetics and correct scoliotic posture; 2) stabilize the spine and stop the progression of the curve; 3) inform patients and their families about the condition and available treatments; 4) enhance breathing; 5) increase activity, including daily living activities and functional mobility; 6) enhance general self-image and self-esteem; and 7) reduce pain. The initial ideas serve as the foundation for BSPTS correctional Principles (Berdishevsky et al 2016).
  Arms: group (2)

SUMMARY:
Adolescent idiopathic scoliosis AIS is the usual diagnosis made in healthy children with a spinal curvature of unknown cause of least 10 degrees but less than 50 degrees. The primary aim of scoliosis management is to stop curvature progression. Anecdotally, the American Academy of Orthopedic Surgeons agree that PSSEs are often considered to produce just as successful of a patient outcome as does surgery.

SEAS has been described as a scoliosis-specific active self-correction technique performed without any external aids and incorporated into functional exercises, The primary goals of SEAS include enhanced posture control, posture rehabilitation, muscle endurance, spinal stability, self-correction, and development of balance stability. Treatment sessions are conducted at least twice a week for 40 minutes each.

Barcelona Scoliosis Physical Therapy School BSPTS method: based on the principles developed by Katharina Schroth, and is mainly used to treat patients with adolescent idiopathic scoliosis, some forms of congenital anteroposterior scoliosis deformities and such other as Scheuermann disease. The predecessor of BSPTS was founded in 1968 in Barcelona, Spain by physiotherapist Elena Salvá. It is a physiotherapy method that includes cognitive, sensory and kinesthetic retraining to improve scoliosis at a three dimensional level. All principles follow a complete posture correction pattern including the trunk, upper and lower limbs. High-intensity forces are applied to the exercises through isometric contractions, stretching and breathing exercises. In summary, the principles of the BSPTS Method as they appear in the international literature are: 3D postural correction, translation, rotation, sagittal expansions, Expansion / Contraction, Stabilization, Integration.

Studies have shown that the BSPTS methodology is also effective in stabilizing the progression of scoliosis. In a one-year study by Zapata and co-authors, the BSPTS group showed effective stabilization of the Cobb angle compared to the observation group.

There isn't any previous study comparing between effect of SEAS approach and BSPTS in treating AIS.

DETAILED DESCRIPTION:
Scoliosis is a three-dimensional spinal abnormality. The most prevalent form of scoliosis is adolescent idiopathic scoliosis AIS. Usually between the ages of 10 and 16. The majority of patients frequently report the first sign of spinal rotation. The thoracic cage's asymmetry and uneven shoulder height follow, along with other abnormalities like razor back, pelvic tilt, falling height, and uneven lower limb length. In extreme situations, movement imbalance and cardiopulmonary dysfunction may also arise. Additionally, because of changes in their physical appearance brought on by the condition, people with AIS may face psychological problems, such as feelings of inadequacy and the possible emergence of psychological disorders. AIS is now a well-known condition that hinders development and growth.

After ruling out all other possible causes of scoliosis, idiopathic scoliosis is determined. Only 0.3% to 0.5% of adolescents with adolescent idiopathic scoliosis AIS, which affects 2% to 3% of the population, will have a curvature of greater than 20 degrees, the magnitude of the curve at which treatment is typically advised. The risk of advancement is highest at the onset of puberty. According to the Heuter-Volkmann principle loading affects vertebral development. In order to better develop conservative treatment for spinal deformity it's better to start during the adolescent growth.

A thorough treatment plan is necessary for the conservative therapy of idiopathic scoliosis because of its complex pathomechanism. Using physiotherapeutic scoliosis-specific exercises PSSE is one of the best ways to address scoliosis. For all schools and techniques that have been approved by the SOSORT, the phrase physiotherapeutic scoliosis-specific exercises PSSE is used. Every approach and school shares a common goal and applies the SOSORT guidelines' tenets. Scientific evidence must serve as the foundation for a PSSE physiotherapy approach that is tailored to each patient. According to the SOSORT consensus, 3D self-correction ranks top among the crucial components that should be incorporated into the exercises . Self-correction is the process by which a patient looks for the optimal alignment they may attain in the three spatial planes.

The BSPTS is the physiotherapy method integrated into the rehabilitation approach used in the 'Elena Salva Institute' in Barcelona, Spain. BSPTS is physiotherapy method that can be defined as a therapy plan of cognitive, sensory-motor and kinaesthetic training which teaches the patient to improve her/his scoliosis posture and soft tissue imbalance, utilizing the assumption that scoliosis posture and soft tissue imbalance promote curve progression. The BSPTS recognizes the importance of multidisciplinary team approach to treat scoliosis which should include medical doctor, physiotherapist, orthotist and psychologist.

The SEAS approach originates from Lyon, some of the base characteristics previously published for the Lyon approach have been retained in SEAS: increasing patient's awareness of the deformity, emphasizing an independent auto-correction by the patient, use of exercises in which balance reactions are elicited. The most important differences gradually developed by SEAS, that made it different from the Lyon approach, include: active three-dimensional self-correction instead of the former auto-elongation, spinal stabilization concept according to the actual physiotherapeutic literature, research of an automatic correct reflex response, namely, a subconscious self-correction which should help to obtain the better integration in the daily life. focus on the cognitive-behavioral approach of the patient to increase compliance to treatment, variability of exercises stimuli instead of absolute repetitive precision of movements, according to modern neurophysiologic knowledge.

Self-correction can be defined as the search for the best possible alignment the patient can achieve in the three spatial planes. Three-dimensional self-correction is considered one of the most important elements for the organization of conservative treatment. The SOSORT (International Society on Scoliosis Orthopedic and Rehabilitation Treatment) consensus in 2005 attributes to the "3D Self-correction" first place in the ranking of important elements to be included in the exercises, The goal of SEAS exercises is to develop an automatic reaction to reaching a more appropriate posture which will encourage the maintenance of a three-dimensionally corrected posture while engaging in daily activities.

ELIGIBILITY:
Inclusion Criteria:

* angle of scoliosis < 30,
* Risser sign of 0-3,
* not participating in other treatment during study
* not using braces.

Exclusion Criteria:

* scoliosis due to congenital, neuromuscular, or syndromic etiology,
* true leg length discrepancy,
* cardiac anomalies, kyphosis, asthma, and other pulmonary diseases.

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-11-01 (Actual)

PRIMARY OUTCOMES:
change of cobbs angle | after 6 months of treatment
  by x-ray assessment of cobbs angle to know the change of the scoliosis curvature
change of sagittal and coronal imbalance | after 6 months of treatment
  laser line machine will be used to assess changes of imbalance of sagittal and coronal
changes of angle of trunk rotation | after 6 months of treatment
  scoliometer is used to assess angle of trunk rotation

SECONDARY OUTCOMES:
assess quality of life | after 6 months of treatment
  SRS-22r patient Questionnaire used to assess quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Bedair Ebrahim, professor of physical therapy, Principal Investigator — kafr-elsheikh university
Locations (1):
- Huda Mohamed Hashad, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No